CLINICAL TRIAL: NCT01888224
Title: Open Label, Balanced, Randomized, Two-treatment, Two-period, Two Sequence, Single Dose, Crossover, Oral Bioequivalence Study of Isotretinoin Capsules 40 mg of Dr. Reddy's Laboratories Limited, India Comparing With Amnesteem Capsules 40 mg of Mylan Pharmaceuticals Inc., in Healthy, Adult, Male Human Subjects Under Fed Conditions.
Brief Title: Bioavailability Study of Isotretinoin Capsules 40 mg Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 618-10
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2011-08

CONDITIONS: Healthy
MeSH Terms: interventions — Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isotretinoin capsules, 40 mg (Experimental): Isotretinoin Capsules, 40 mg of Dr.Reddy's Laboratories Ltd
  Interventions: Drug: Isotretinoin
- AMNESTEEM (Active Comparator): AMNESTEEM 40 mg of Mylan Pharmaceuticals Inc
  Interventions: Drug: Isotretinoin

INTERVENTIONS:
Drug: Isotretinoin — Isotretinoin Capsules,40 mg
  Other Names: AMNESTEEM

SUMMARY:
To characterise the pharmacokinetic profile of sponsor's test formulation Isotretinoin Capsules 40 mg in comparison to the reference formulation Amnesteem (Containing Isotretinoin) Capsules 40 mg after single oral dose administration to healthy, normal, adult, human male subjects under fed condition.

DETAILED DESCRIPTION:
An open label, balanced, randomized, two-treatment, two-period, two sequence, single dose, crossover, oral bioequivalence study of Isotretinoin Capsules 40 mg under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult human male volunteers between 18 to 45 years of age (both inclusive) living in and around Ahmedabad city or western part of India.
* Having a Body Mass Index (BMI) between 18.5-27.5 (both inclusive), calculated as weight in kg / height in meter2.
* Not having any significant disease in medical history or clinically significant abnormal findings during screening, medical history, physical examination,laboratory evaluations, 12- lead ECG and X-ray chest recordings.
* Able to understand and comply with the study procedures, in the opinion of the principal investigator.
* Able to comply to use 2 forms of effective contraception methods simultaneously during Isotretinoin study, and for 1 month after study.
* Able to give voluntary written informed consent for participation in the trial.
* Able to read and/or understand drug medication Guide either in English or in a provided translation when given along with informed consent form.

Exclusion Criteria

* Known hypersensitivity or idiosyncratic reaction to Isotretinoin or any of the excipients including parabens or any related drug.
* History or presence of any disease or condition which might compromise the haemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system.
* Ingestion of any medicine including herbal medicines at any time within 14 days before dosing in Period I. In any such case subject selection will be at the discretion of the Principal Investigator.
* Any history or presence of asthma (including aspirin induced asthma) or nasal polyp or NSAID induced urticaria.
* Use of any recreational drugs or history of drug addiction or testing positive in prestudy drug scans.
* A recent history of harmful use of alcohol(less than 2 years), i.e. alcohol consumption of more than 14 standard drinks per week (A standard drink is defined as 360 ml of beer or 150 ml of wine or 45 ml of 40% distilled spirits, such as rum,whisky, brandy etc) or consumption of alcohol or alcoholic products within 48 hours prior to receiving study medicine.
* Smokers, who smoke 10 or more than 10 cigarettes / day or inability to abstain from smoking during the study.
* The presence of clinically significant abnormal laboratory values during screening.
* History or presence of psychiatric disorders.
* A history of difficulty in donating blood.
* Donation of blood (1 unit or 350 mL) or receipt of an investigational medicinal product or participation in a drug research study within a period of 90 days prior to the first dose of study medication. Elimination half-life of the study drug should be taken into consideration for inclusion of the subject in the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2011-06; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) | Pre-dose (0) and 0.5, 1,1.5,2,2.5,3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8,10,12,16,20,24, 36, 48,72 and 96 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Alpeshkumar Patel, MD, Principal Investigator — Lambda Therapeutic Research Limited
Locations (1):
- Lambda Therapeutic Research Ltd.,, Ahmedabad, Gujarat, India